CLINICAL TRIAL: NCT02985983
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Study With an Open Label Extension to Evaluate the Efficacy and Safety of Brodalumab in Subjects With Axial Spondyloarthritis
Brief Title: A Study of Brodalumab in Subjects With Axial Spondyloarthritis (axSpA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4827-006
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Axial Spondyloarthritis
Keywords: Brodalumab; Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brodalumab (Experimental): Brodalumab administered SC
  Interventions: Drug: Brodalumab
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brodalumab — Administered Brodalumab by subcutaneous (SC) injection until week 66.
  Arms: Brodalumab
Drug: Placebo — Administered Placebo by subcutaneous (SC) injection until week 16. Administered Brodalumab by SC injection from week 17 until week 66.
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of Brodalumab in axSpA (ankylosing spondylitis [AS] and non-radiographic axial spondyloarthritis [nr-axSpA]) subjects compared to placebo, as measured by the proportion of axSpA subjects achieving an Assessment of SpondyloArthritis international Society (ASAS) 40 response at week 16.

ELIGIBILITY:
Inclusion Criteria:

* Subject with age at onset <45 years and continuous chronic back pain for ≥ 3 months fulfills the ASAS classification criteria of axial spondyloarthritis (with the exception of the Crohn's disease)
* Subject has Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score ≥ 4 at screening and enrollment
* Subject has spinal pain score (BASDAI question #2) ≥ 4 at screening and enrollment
* Subject has had adequate therapy with non-steroidal anti-inflammatory drugs (oral NSAIDs) for back pain for at least 3 months with inadequate treatment response before enrollment

Exclusion Criteria:

* Complete ankylosis (fusion) of the spine
* Subject with active ongoing inflammatory diseases other than axSpA that might confound the evaluation of Brodalumab therapy, including reactive arthritis, spondyloarthritis associated with inflammatory bowel disease, SAPHO syndrome (pustulotic arthro-osteitis), fibromyalgia, ankylosing spinal hyperostosis, osteitis condensans ilii, spondylosis deformans, or osteoarthritis sacroiliac joint disease
* Subject has a prior history of >1 anti-tumor necrosis factor (TNF) therapy
* Subject has a history or evidence of suicidal ideation (severity of 4 or 5) or any suicidal behavior based on an assessment with the Columbia-Suicide Severity Rating Scale (C-SSRS) at enrollment
* Subject has a history or evidence of a psychiatric disorder, alcohol and/or substance abuse
* Subject has severe depression based on a total score of ≥ 15 on the Patient Health Questionnaire-8 (PHQ-8) at enrollment (note: subjects with a total score of 10 to 14 on the PHQ-8 should be referred to a mental health care professional)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Percentage of ASAS 40 in axSpA subjects | Week 16

SECONDARY OUTCOMES:
Percentage of ASAS 40 in AS subjects | Week 16
Percentage of ASAS 40 in nr-axSpA subjects | Week 16
Ankylosing Spondylitis Disease Activity Score (ASDAS)-CRP change from baseline in axSpA subjects | Week 16
Number of adverse events | Up to week 68
Number of patients exposed to anti-KHK4827 antibodies | Pre-dose,Week 16,Week 32,Week 48,Week 68 or End of study
Serum KHK4827 concentration | pre-dose、Week 1、Week 2、Week 4、Week 8、Week 12、Week 14、Week 16、Week 24、Week 28、Week 32

CONTACTS AND LOCATIONS:
Locations (48):
- Japan (25):
  - Fujita Health University Hpspital, Aichi
  - Tokyo Women's Medical University Yachiyo Medical Center, Chiba
  - Chihaya Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Kyusyu University Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Katayama Seikeigeka Rheumatism Clinic, Hokkaido
  - Hyogo College of Medicine, Hyōgo
  - Kagawa University Hospital, Kagawa
  - Kochi Medical School Hospital, Kochi
  - Sasebo Chuo Hospital, Nagasaki
  - Tenri Hospital, Nara
  - Okayama Saiseikai Outpatient Centerl Hospital, Okayama
  - Okinawa Prefectural Chubu Hospital, Okinawa
  - Tomishiro Central Hospital, Okinawa
  - National Hosptal Organization Osaka Minami Medical Center, Osaka
  - Osaka City General Hospital, Osaka
  - Osaka City University Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Yukioka Hospital, Osaka
  - Juntendo University Hospital, Tokyo
  - St.Luke's International Hospital, Tokyo
  - Toho University Ohashi Medical Center, Tokyo
  - Toho University Omori Medical Center, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
- South Korea (12):
  - Pusan National University Hospital, Busan
  - Daegu Catholic University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Ajou University Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - KyungHee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The catholic university of korea Seoul St.mary's Hospital, Seoul
- Taiwan (11):
  - Chang Gung Medical Foundation, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Cathay General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation, LinKou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim TH, Kishimoto M, Wei JC, Jeong H, Nozaki A, Kobayashi S. Brodalumab, an anti-interleukin-17 receptor A monoclonal antibody, in axial spondyloarthritis: 68-week results from a phase 3 study. Rheumatology (Oxford). 2023 May 2;62(5):1851-1859. doi: 10.1093/rheumatology/keac522. PMID 36130275
- [Derived] Wei JC, Kim TH, Kishimoto M, Ogusu N, Jeong H, Kobayashi S; 4827-006 study group. Efficacy and safety of brodalumab, an anti-IL17RA monoclonal antibody, in patients with axial spondyloarthritis: 16-week results from a randomised, placebo-controlled, phase 3 trial. Ann Rheum Dis. 2021 Aug;80(8):1014-1021. doi: 10.1136/annrheumdis-2020-219406. Epub 2021 Apr 7. PMID 33827787